CLINICAL TRIAL: NCT01608347
Title: Low Molecular Weight Heparin for Treatment of Recurrent Miscarriage With Negative Antiphospholipid Antibodies: a Randomized Controlled Trial
Brief Title: Low Molecular Weight Heparin in Recurrent Miscarriage With Negative Antiphospholipid Antibodies
Acronym: LMWH-APAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Omar Mamdouh Shaaban (Other)
Responsible Party: Sponsor-Investigator, Omar Mamdouh Shaaban, Dr, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAPAN
Record Dates: First submitted 2012-05-26; First posted 2012-05-31 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Recurrent Miscarriage
Keywords: LMWH; enoxaparin; recurrent miscarriage; continuing fetal viability beyond 20 weeks gestation
MeSH Terms: conditions — Abortion, Habitual | interventions — Enoxaparin; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LMWH + Folic acid group (Experimental): Daily 40 mg of enoxaparin (LMWH) (Clexane, Sanofi Aventis, Paris, France)subconsciously started once positive pregnancy test. Treatment will be continued until abortion or delivery (if premature), or 37 weeks of pregnancy. Additionally, 500 micrograms Folic acid tab once/daily until 13 weeks' of gestation.
  Interventions: Drug: LMWH+Folic acid
- Folic acid (Active Comparator): 500 microgram folic acid tab/day started once positive pregnancy test and will be continued until 13 weeks' of gestation.
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Drug: LMWH+Folic acid — Patients will receive a fixed dose of 40 mg of enoxaparin subcutaneous daily. Treatment will start once positive pregnancy test and will be continued until abortion or delivery (if premature), or 37 weeks of pregnancy. Additionally, 500 micrograms Folic acid tablet once daily will be started once positive pregnancy test and continues until 13 weeks' of gestation.
  Other Names: (Clexane, Sanofi Aventis, Paris, France)
  Arms: LMWH + Folic acid group
Drug: Folic Acid — Folic acid 500 micrograms daily once positive pregnancy test until the 13th week of pregnancy or abortion
  Arms: Folic acid

SUMMARY:
Recurrent miscarriage (RM) is traditionally defined as three or more consecutive miscarriages occurring before 20 weeks post-menstruation. It is one of the most common clinical problems in reproduction, yet a definite cause can be established in only 50 percent of cases (ACOG practice bulletin, 2002). Many etiological factors have been proposed but none of them has been fully substantiated. RM has been directly associated with maternal thrombophilic disorders, parental chromosomal anomalies, and structural uterine anomalies and indirectly with maternal immune dysfunction and endocrine abnormalities.

The association between pregnancy loss and antiphospholipid antibodies (aPL) was first noticed in the latter third of the last century. The antiphospholipid syndrome (APS) is characterized by the presence of antiphospholipid antibodies (APLA), associated with venous and/or arterial thrombosis, and/or pregnancy loss. The adverse pregnancy outcomes associated with the presence of APLAs include: recurrent fetal loss, intrauterine growth restriction (IUGR), and severe pre-eclampsia especially of early onset.

Testing the effect of Heparin in treatment of cases with RA but negative for APA has bee done in few animal and clinical studies. Animal studies showed that the subset of cases with disorders suspicious for APS but who had negative test results for LAC and aCL is carrying antibodies pathogenic to murine pregnancy. Testing other immunoglobulin G may provide additional means to identify cases with an yet uncharacterized immune condition. Moreover, the clinical relevance of low levels of APLA in these women remains unproved.

Randomized prospective study was done to assess the efficacy of early thromboprophylaxis of Low molecular weight heparin (LMWH) (Enoxaparin sodium 20 mg, once daily subcutaneously) in women with a history of recurrent miscarriages without identifiable causes versus no treatment. The results showed that, there is a significant reduction in the incidence of both early and late miscarriages (8.8% vs 4.1%) (2.3% versus 1.1%) with or without treatment, respectively.

Cochrane Database systemic review (2005) shows randomized comparative studies for treating recurrent miscarriage in women without antiphospholipid syndrome. The first group treated by low dose aspirin alone and the second group treated by low dose aspirin + LMWH. The result of these studies shows that no significant differences between the two groups and identify the need of large randomized controlled trial to solve this problem.

The above evidence suggests the probability of presence of untested LAC and aCL or very low levels of APLA by commonly used methods in women with recurrent miscarriage. These antibodies may explain recurrent miscarriage in cases with negative antiphospholipid antibodies. It remains to test the efficacy of heparin (proven effective treatment in those with positive antibodies) in the patients with negative antibodies. Finding a solution to this frustrating problem may open the way for an unsolved problem.

The proposed study is an open labeled randomized controlled trial (RCT) To evaluate the effect of LMWH versus no heparin in treatment of recurrent miscarriage that is negative for antiphospholipid antibodies testing.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between 20-35 years of age with a history of regular marital life with the same partner.
2. Had at least 3 previous consecutive pregnancy losses before 20 weeks of gestation.
3. Regularly menstruating before current pregnancy.
4. Got spontaneous conception.
5. Negative antibody tests for antiphospholipid syndrome. IgG and IgM aCL antibodies will be detected by an enzyme linked immunoabsorbent assay (ELISA. The results considered positive when the IgG aCL > 8.4 IU/ml; IgM aCL > 7 IU/ml.

Exclusion Criteria:

1. Presence of polycystic ovarian syndrome which diagnosed either by history suggestive or PCO appearance by TV Ultrasonography.
2. Abnormal uterine cavity as proved by sonohysterography or diagnostic hysteroscopy.
3. Positive consanguinity between the two partners.
4. Presence of any other endocrine abnormalities. Glucose tolerance curve will be done exclude the presence of diabetes. Other endocrine abnormalities will be excluded by history and clinical examination. If any clinical suspicion has been raised, the required endocrinological tests will be done.
5. Women refused to participate in the trial.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Continuation of viable pregnancy beyond 20 weeks gestation | 20 weeks gestation
  Number of patients who will continue with a viable pregnancy beyond 20 weeks gestation

SECONDARY OUTCOMES:
Fetal viability at the end of the 34th week of pregnancy. | 34 weeks gestation
Normal fetal anatomy by ultrasound scan | 20 weeks gestation
Side effect encountered from treatment | 20 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Omar M SHaaban, MD, Principal Investigator — Assiut University